CLINICAL TRIAL: NCT05964738
Title: Safety and Tolerability of Diuretics Withdrawal in Heart Failure with Reduced Ejection Fraction. REDICAE Trial.
Brief Title: Effect of Diuretics Withdrawal in Chronic Heart Failure with Reduced Ejection Fraction
Acronym: REDICAE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Sociedad Andaluza de Cardiología (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REDICAE
Record Dates: First submitted 2023-06-28; First posted 2023-07-28 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Electric Impedance; Dyspnea; Safety; Withdrawal
Keywords: Heart Failure; Diuretics; Dyspnea; Safety; Fluid overload; Withdraw; Electric Impedance
MeSH Terms: conditions — Heart Failure; Dyspnea; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diuretics withdrawal (Experimental)
  Interventions: Drug: Diuretics withdrawal
- Diuretics maintenance (Active Comparator)
  Interventions: Drug: Diuretics maintenance

INTERVENTIONS:
Drug: Diuretics withdrawal — Diuretics that not have been demonstrated improve survival in chronic HFrEF are withdrawn
  Arms: Diuretics withdrawal
Drug: Diuretics maintenance — Any diuretic could be used
  Arms: Diuretics maintenance

SUMMARY:
REDICAE trial was designed to evaluate the safety and tolerability of diuretics withdrawal in stable, euvolemic chronic outpatients with heart failure with reduced ejection fraction. It is a single-center, randomized, open-label, phase II clinical trial.

DETAILED DESCRIPTION:
Treatment of heart failure with reduced ejection fraction (HFrEF) has improved patient survival in recent decades. Diuretics are essentials in acute decompensated heart failure, specially furosemide. However, when patients are stable and euvolemic diuretics (loop diuretics, thiazide diuretics or acetazolamide) might increase adverse effects: renin-angiotensin-aldosterone system activation, renal function impairment or electrolyte disturbances.

The 2021 European Society of Cardiology (ESC) Guidelines for the diagnosis and treatment of acute and chronic heart failure recommend angiotensin-converting enzyme inhibitors (ACEI) or angiotensin receptor-neprilysin inhibitor (ARNI), beta-blockers (BB), mineralocorticoid receptor antagonists (MRA) and sodium-glucose co-transporter 2 inhibitors (iSTLT2) as first-line therapy for HFrEF. A significant proportion of patients take a maintenance diuretics dose despite the clinical benefits and prognosis are controversial.

Current clinical guidelines suggest that diuretic use can be reduced or discontinued in selected euvolemic or hypovolemic patients. This statement is based on the results of the ReBIC-1 trial published in 2019, which showed a neutral effect of furosemide discontinuation in stable chronic outpatients with HFrEF treated according to the 2016 ESC heart failure guidelines standards of care.

REDICAE trial was designed to evaluate the safety and tolerability of diuretics withdrawal, not just furosemide, in stable euvolemic chronic outpatients with HFrEF. It is a single-center, randomized, open-label phase II clinical trial.

The pathophysiology of congestion in heart failure is complex and multifactorial. In the REDICAE trial, volume status will be determined by biomarkers, echocardiography and bioelectrical impedance analysis. The patients enrolled in the study will be under contemporary guideline-directed medical therapy, including SGLT2 inhibitors. This trial is the largest prospective trial evaluating the clinical effects of diuretic discontinuation in HFrEF patients under contemporary pharmacological therapy for heart failure.

REDICAE trial develops in Hospital Universitario Reina Sofía in Cordoba (Spain)

ELIGIBILITY:
INCLUSION CRITERIA:

* Outpatients diagnosed of chronic HFrEF by criteria of ESC Guidelines of 2021
* Age equal or greater than 18 year-old
* Stable and euvolemic outpatients determined by clinical criteria, biomarkers (CA-125 < 23 U/mL) and bioelectrical impedance analysis
* Left Ventricular Ejection Fraction less than 50% by echocardiography or cardiovascular magnetic resonance performed within 6 months before the screening visit
* New York Heart Association functional class I or II
* No episodes of acute decompensated heart failure within 2 months before the screening visit
* Treatment with a stable dose of diuretic for at least 1 month before the screening visit
* Optimal medical therapy with ACEI/ARNI, BB, MRA and iSGLT2 must be started to titration unless any of them were contraindicated or not tolerated
* Plasma potassium < 5 mg/dl in the screening visit

EXCLUSION CRITERIA:

* Acute coronary syndrome within 3 months before screening visit
* Awaiting cardiac resynchronization therapy
* Any severe valve heart disease not yet treated
* Pulmonary hypertension or any severe pulmonary disease
* End-stage chronic kidney disease (on hemodialysis). Acute kidney injury
* Severe hepatic failure or cirrhosis
* Malignancy on active treatment
* Congenital heart disease
* Awaiting cardiac transplantation
* Inability to understand and sign the informed consent
* Participation in any other interventional clinical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Dyspnea assessed by a visual analogue scale (VAS) | baseline - 30 days - 90 days - 180 days
  VAS scores are scaled from 0 to 100 millimeters (mm). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Acute decompensated heart failure events | 180 days
  Number of Hospital admissions, emergency department visits or unscheduled medical appointments requiring intravenous diuretic treatment, and increase in diuretic dose or reintroduction of an oral diuretic.
Variation of plasmatic levels of natriuretic peptides | baseline - 30 days - 90 days - 180 days
  Levels of the N-terminal pro b-type natriuretic peptide (NT-proBNP)
Tissue fluid overload | baseline - 30 days - 90 days - 180 days
  Variation of plasmatic levels of antigen carbohydrate 125 (CA-125)
Body Composition Monitor (BCM) of Fresenius Medical Care | baseline - 30 days - 90 days - 180 days
  Variation of fluid overload assessed by bioelectrical impedance analysis
Inferior vena cava (IVC) diameter | baseline - 30 days - 90 days - 180 days
  IVC diameter measured in its intra-hepatic portion at 2 cm of the junction with the hepatic veins using a longitudinal view from a sub-xiphoid position. IVC is dilated when its diameter is more than 20 mm.
Hepatic vein Doppler | baseline - 30 days - 90 days - 180 days
  Pulsed wave Doppler shows a systolic (S) and diastolic (D) components. Normal pattern (S > D), mildly abnormal pattern (S < D) and severely abnormal pattern (S reverses)
Portal vein Doppler | baseline - 30 days - 90 days - 180 days
  Pulsed wave Doppler shows a continuous nonpulsatile flow. Using the pulsatility fraction (PF=100*[(Vmax - Vmin)/Vmax)]) are three patterns: normal PF < 30%, mildly abnormal PF 30-50% and severely abnormal PF >50%.
Intra-renal venous Doppler | baseline - 30 days - 90 days - 180 days
  Pulsed wave Doppler shows a normal pattern when flow is continuous. Mildly abnormal pattern shows a biphasic flow (S and D). Severely abnormal pattern shows a monophasic flow (D)
Ultrasound congestion parameters by Venous Excess Ultrasound (VExUS) protocol | baseline - 30 days - 90 days - 180 days
  IVC diameter, hepatic vein Doppler, portal vein Doppler and intra-renal venous Doppler patterns are combined to report VExUS grades:
  * Grade 0 (no congestion): IVC < 20 mm
  * Grade 1 (mild congestion): IVC ≥ 20 mm and any combination of normal or mildly abnormal pattern
  * Grade 2 (moderate congestion): IVC ≥ 20 mm + ≥ 1 severely abnormal pattern
  * Grado 4 (severe congestion): IVC ≥ 20 mm + ≥ 2 severely abnormal pattern
Congestion assessed by lung ultrasound | baseline - 30 days - 90 days - 180 days
  Pleural effusion or pathological B lines. More than two B lines are considered as pathological.
Quality of life status | baseline - 30 days - 90 days - 180 days
  Change From Baseline in the Kansas City Cardiomyopathy Questionnaire 12 (KCCQ-12) score. KCCQ-12 scores are scaled from 0 to 100. Higher scores mean a better outcome.
6 minute walk test | baseline - 30 days - 90 days - 180 days
  Change From Baseline in meters walked, as assessed by the 6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Torres Zamudio, MD, Principal Investigator — Hospital Universitario Reina Sofía de Córdoba; Juan Carlos Castillo Domínguez, MD, PhD, Study Director — Maimónides Biomedical Research Institute of Córdoba
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Córdoba (Andalucía), Spain

IPD SHARING:
Plan to Share IPD: Yes
Contact by email with Central Contact Person
Supporting Information: Study Protocol, ICF, CSR
Time Frame: From October 2024
Access Criteria: Contact by email with Central Contact Person

REFERENCES:
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Vardeny O, Claggett B, Kachadourian J, Desai AS, Packer M, Rouleau J, Zile MR, Swedberg K, Lefkowitz M, Shi V, McMurray JJV, Solomon SD. Reduced loop diuretic use in patients taking sacubitril/valsartan compared with enalapril: the PARADIGM-HF trial. Eur J Heart Fail. 2019 Mar;21(3):337-341. doi: 10.1002/ejhf.1402. Epub 2019 Feb 11. PMID 30741494
- [Background] Jackson AM, Dewan P, Anand IS, Belohlavek J, Bengtsson O, de Boer RA, Bohm M, Boulton DW, Chopra VK, DeMets DL, Docherty KF, Dukat A, Greasley PJ, Howlett JG, Inzucchi SE, Katova T, Kober L, Kosiborod MN, Langkilde AM, Lindholm D, Ljungman CEA, Martinez FA, O'Meara E, Sabatine MS, Sjostrand M, Solomon SD, Tereshchenko S, Verma S, Jhund PS, McMurray JJV. Dapagliflozin and Diuretic Use in Patients With Heart Failure and Reduced Ejection Fraction in DAPA-HF. Circulation. 2020 Sep 15;142(11):1040-1054. doi: 10.1161/CIRCULATIONAHA.120.047077. Epub 2020 Jul 16. PMID 32673497
- [Background] Packer M, Anker SD, Butler J, Filippatos G, Ferreira JP, Pocock SJ, Sattar N, Brueckmann M, Jamal W, Cotton D, Iwata T, Zannad F; EMPEROR-Reduced Trial Committees and Investigators. Empagliflozin in Patients With Heart Failure, Reduced Ejection Fraction, and Volume Overload: EMPEROR-Reduced Trial. J Am Coll Cardiol. 2021 Mar 23;77(11):1381-1392. doi: 10.1016/j.jacc.2021.01.033. PMID 33736819
- [Background] Rohde LE, Rover MM, Figueiredo Neto JA, Danzmann LC, Bertoldi EG, Simoes MV, Silvestre OM, Ribeiro ALP, Moura LZ, Beck-da-Silva L, Prado D, Sant'Anna RT, Bridi LH, Zimerman A, Raupp da Rosa P, Biolo A. Short-term diuretic withdrawal in stable outpatients with mild heart failure and no fluid retention receiving optimal therapy: a double-blind, multicentre, randomized trial. Eur Heart J. 2019 Nov 21;40(44):3605-3612. doi: 10.1093/eurheartj/ehz554. PMID 31424503
- [Background] Romano G, Vitale G, Bellavia D, Agnese V, Clemenza F. Is diuretic withdrawal safe in patients with heart failure and reduced ejection fraction? A retrospective analysis of our outpatient cohort. Eur J Intern Med. 2017 Jul;42:e11-e13. doi: 10.1016/j.ejim.2017.03.025. Epub 2017 Apr 6. No abstract available. PMID 28390780
- [Background] Nunez J, Bayes-Genis A, Revuelta-Lopez E, Ter Maaten JM, Minana G, Barallat J, Cserkoova A, Bodi V, Fernandez-Cisnal A, Nunez E, Sanchis J, Lang C, Ng LL, Metra M, Voors AA. Clinical Role of CA125 in Worsening Heart Failure: A BIOSTAT-CHF Study Subanalysis. JACC Heart Fail. 2020 May;8(5):386-397. doi: 10.1016/j.jchf.2019.12.005. Epub 2020 Mar 11. PMID 32171764
- [Background] Ekman I, Granger B, Swedberg K, Stenlund H, Boman K. Measuring shortness of breath in heart failure (SOB-HF): development and validation of a new dyspnoea assessment tool. Eur J Heart Fail. 2011 Aug;13(8):838-45. doi: 10.1093/eurjhf/hfr062. PMID 21791539